CLINICAL TRIAL: NCT06467162
Title: The Usage of Spacers and the Relationship With Symptoms Severity in Chronic Obstructive Pulmonary Disease Elderly Patients: A Correlational Study
Brief Title: Usage of Spacers and the Relationship With Symptoms Severity in COPD Elderly Patients
Status: Completed | Type: Observational
Sponsor: Ai-Ling Chang (Other)
Responsible Party: Sponsor-Investigator, Ai-Ling Chang, Supervisor, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Other Study IDs: 1110206
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Disease; Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease; Spacer; Symptom severity
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: Research participants were interviewed using structured questionnaires, including demographic characteristics information, clinical characteristics information, and the chronic obstructive pulmonary disease assessment test.

SUMMARY:
The goal of this observational study is to investigate the usage of spacers and their relationship with symptom severity in chronic obstructive pulmonary disease elderly patients. Patients with chronic obstructive pulmonary disease aged 65 years or over at thoracic medicine outpatient clinics were recruited in this study. Research participants were interviewed using structured questionnaires, including demographic characteristics information, clinical characteristics information, and the chronic obstructive pulmonary disease assessment test.

DETAILED DESCRIPTION:
The goal of this observational study is to investigate the usage of spacers and their relationship with symptom severity in chronic obstructive pulmonary disease elderly patients. A convenience sample was used to recruit patients with chronic obstructive pulmonary disease aged 65 years or over at thoracic medicine outpatient clinics from a teaching hospital in Taiwan. Research participants were interviewed using structured questionnaires, including demographic characteristics information, clinical characteristics information, and the chronic obstructive pulmonary disease assessment test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 or above diagnosed with COPD by a pulmonologist.
* Clear consciousness and communication abilities in Mandarin or Taiwanese.
* Consent to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients who are blind, deaf, unable to express themselves, and unable to understand the study explanation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with chronic obstructive pulmonary disease aged 65 years or over at thoracic medicine outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Symptoms severity | Immediately after the outpatient department visit
  The severity and impacts of the COPD symptoms were measured by using the chronic obstructive pulmonary disease assessment test

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ting Huang, PhD, Study Chair — Da-Yeh University
Locations (1):
- Wan-Ting Huang, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No